CLINICAL TRIAL: NCT04231890
Title: Early Identification and Prevention of Extubation Failure in Adults Using Integrated Pulmonary Index: A Randomized Controlled Trial
Brief Title: Early Identification and Prevention of Extubation Failure in Adults Using Integrated Pulmonary Index
Acronym: IPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Ramandeep Kaur, Research Coordinator; MSc, RRT-ACCS, AE-C, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 18112803
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Mechanical Ventilation Complication; Extubation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPI group (Experimental): IPI monitoring
  Interventions: Other: IPI monitoring
- Control group (No Intervention): Standard monitoring

INTERVENTIONS:
Other: IPI monitoring — Patients in this arm will have IPI monitoring
  Arms: IPI group

SUMMARY:
The primary aim of this study is to compare reintubation rate when using standard medical therapy (SMT) versus a monitoring tool, Integrated Pulmonary Index (IPI), to alert clinicians of the patient's respiratory status and need for therapy after planned extubation.

DETAILED DESCRIPTION:
The study is designed as a randomized controlled trial to compare two methods to guide application of clinical interventions after planned extubation: SMT versus IPI based clinical management among adult patients admitted in the ICU and receiving mechanical ventilation for ≥24 hours. Each mechanically ventilated subject within the inclusion criteria and with a physician order for extubation will be randomized to either the SMT or IPI based clinical management group. Once the extubation order is placed by the medical team, the patient will be randomized to IPI monitoring group or standard medical management group. Patients randomized to IPI group will be placed on IPI monitoring after extubation.Respiratory Therapist (RT) will extubate and connects the patient to EtCO2 cannula (Medtronic, Minneapolis, MN) and will turn on IPI monitoring on the Philips monitor. Any subject with decrease in IPI by 1 within 1 hour of extubation or IPI ≤ 4 after 1 hour of extubation will be assessed by RT and will receive standard medical therapy based on respiratory department protocols. IPI monitoring will be continued for up to 72 hours after extubation. Patients randomized to control group will receive standard medical therapy based on the respiratory department protocols. All patients will be clinically monitored for 72 hours after extubation to assess the extubation outcome. Patients that require reintubation will be reintubated based on the medical team decision and will be discontinued from the study. Patients that do not require reintubation after 72 hours will successfully complete the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects 18 years and older, endotracheally intubated and receiving assisted mechanical ventilation for more than 24hours, and
* Subjects under planned extubation based on the medical team approval

Exclusion Criteria:

* Subjects who are less than 18 years old,
* are pregnant,
* have tracheostomy tube as they do not qualify for extubation,
* have do-not-resuscitate or do-not-intubate orders,
* accidental or self-extubated patients,
* reintubation after study enrollment,
* are extubated terminally, or
* receiving extracorporeal membrane oxygenation (ECMO)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Reintubation rate at 72hours | 72 hours
  Reintubation rate defined as requiring re-intubation and returning to mechanical ventilation within 72 hours after the initial discontinuation from the ventilation due to respiratory failure

SECONDARY OUTCOMES:
Reintubation rate at 7 days | 7 days
  Reintubation rate defined as requiring re-intubation and returning to mechanical ventilation within 7 days after the initial discontinuation from the ventilation due to respiratory failure
ICU length of stay | upto 12 weeks
  Total ICU day
ICU mortality | upto 12 weeks
  Patient status at the time of ICU discharge

CONTACTS AND LOCATIONS:
Overall Officials: David Vines, PhD, Study Chair — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaur R, Vines DL, Harnois LJ, Elshafei A, Johnson T, Balk RA. Identification and Prevention of Extubation Failure by Using an Automated Continuous Monitoring Alert Versus Standard Care. Respir Care. 2022 Oct;67(10):1282-1290. doi: 10.4187/respcare.09860. Epub 2022 Mar 28. PMID 35347080